CLINICAL TRIAL: NCT03338283
Title: Short-term Efficacy of Interferential Current Electro-massage on Self-perceived Pain and Function in Subjects With Subacromial Pain Syndrome: A Randomized Clinical Trial
Brief Title: Electro-massage in Subjects With Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USBlanca
Record Dates: First submitted 2017-10-29; First posted 2017-11-09 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Subacromial Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromassage (Experimental): Electromassage and conservatory treatment. All subjects will be received a conservatory treatment (1h and 40 min) and electro-massage (10min).
  The protocol will consist of six sessions, twice a week for three weeks. The duration will be 1 hour and 40 min for the conservatory treatment and 10 min for the electro-massage.
  Interventions: Other: Electromassage
- Conservatory Treatment (Active Comparator): The control protocol will combine: (a) thermotherapy with infrared application; (b) active, self-assisted and isometric shoulder exercises, including Codman's pendulum exercises; (c) manual therapy, always in a pain-free range of movement; and (d) ultrasound in pulsatile mode over the acromium and scapulohumeral area.
  Interventions: Other: Conservatory treatment

INTERVENTIONS:
Other: Electromassage — Electro-massage that will be performed by a specialist physiotherapist with more than 8 years of experience We use ENDOMED 482 (Enraf Nonius, Spain) for the elecro-massage. the current parameters are: frequency shift at 4000 Hz IFC, 100 Hz AMF in CV mode. We will gradually raise the current intensity until reaching a high level, but not so high as to cause pain or discomfort, nor evident muscle contraction, although a gentle vibration is allowed. The electro-massage was performed on the musculature of the shoulder and neck.
  Arms: Electromassage
Other: Conservatory treatment — The control protocol will combine: (a) thermotherapy with infrared application; (b) active, self-assisted and isometric shoulder exercises, including Codman's pendulum exercises; (c) manual therapy, always in a pain-free range of movement; and (d) ultrasound in pulsatile mode over the acromium and scapulohumeral area.
  Arms: Conservatory Treatment

SUMMARY:
Objectives: Establishing and validating an electrotherapy procedure with interferential current (IFC) application using electro-massage on patients who have undergone acromioplasty surgery. To evaluate the possible decrease in pain perception and improvement of functionality following surgical intervention.

Design: Randomized, single blind clinical trial. Subjects: 18-patients, aged 18 to 65, with a similar distribution of male and female participants Methods: 10-patients will be enrolled in the experimental group and 8 patients as the control group. Both groups of patients will undergo six physiotherapy sessions (three times a week). The experimental group will undergo a treatment consisting of electro-massage with constant voltage (CV) IFC bipolar application, 4000 Hz carrier current and 100 Hz amplitude modulated frequency (AMF). Two 48 cm2 electrodes will be used. Session length with electrotherapy will be approximately ten minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients having undergone acromioplasty surgery in the three months prior to the first day of Physiotherapy treatment

Exclusion Criteria:

* Value equal to or less than 45 in Personal Psychological Apprehension Scale, showing any absolute contraindication for Physiotherapy or Electrotherapy treatment, fear or apprehension for Electrotherapy application, not signing informed consent, showing alterations in local level sensitivity (cervical-scapulohumeral complex), showing bone fracture associated with SCS, having been applied local infiltration with corticoids following surgery and having started Physiotherapy treatment before signing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Pain level, assessed by Visual Analogue Scale | Change from Baseline Pain level at 3 weeks
  This scale is the most accepted to calculate pain level. The range is from 0 (no pain) to 10 (hard pain).

SECONDARY OUTCOMES:
Functional evaluation, assessed by Constant Scale. Reference: Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4 | Change from Baseline Constant Scale at 3 weeks
  This scale is the most accepted at European level. It calculates pain, activities of daily living, mobility and strength. It is a scale validated by the European Society of Shoulder and Elbow Surgery. Several subscales are combined to compute a total score.

OTHER OUTCOMES:
Range of shoulder´s motion (ROM) | Change from Baseline ROM at 3 weeks
  The flexion, extension, abduction, adduction, internal and external rotation were analyzed. They were measured by goniometer (iPhone app).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Albornoz-Cabello, PhD, Study Director — University of Seville
Locations (1):
- Department of Physiotherapy. Faculty of Nursing, Physiotherapy and Podiatry, Seville, Spain

IPD SHARING:
Plan to Share IPD: No